CLINICAL TRIAL: NCT06806358
Title: Clinical and Ultrasonographic Predictors of IUD Related Complications: A Prospective Cohort Study
Brief Title: Clinical and Ultrasonographic Predictors of IUD Related Complications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N 362
Record Dates: First submitted 2025-01-21; First posted 2025-02-04 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: IUCD Complication

STUDY DESIGN:
Intervention Model Description: IUCD insertion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IUD insertion (Experimental): IUD insertion in women needing contraception
  Interventions: Device: IUD insertion

INTERVENTIONS:
Device: IUD insertion — * Perform a bimanual examination
  * Insert a warm, moistened speculum.
  * Cleanse the cervix with an antiseptic solution.
  * Open the sterile insertion instruments without touching
  * Remove the tenaculum by its handle and grasp the anterior or posterior lip of the cervix.
  * Apply gentle traction with the tenaculum to straighten the canal.
  * Remove the sound by its handle and gently insert it to measure the depth of the uterus. Do not apply great force if there is resistance. Apply further traction to the tenaculum and attempt to re-insert the sound at a different angle. Once the sound is inserted and removed
  * Open the IUD pack without touching its contents.
  * Put on sterile gloves.
  * Load the IUD and insert it into the uterine cavity according to the manufacturer instructions.
  * Gently remove the tenaculum.
  * Trim the strings of the IUD to 3-4 cm in length
  * Remove the speculum and assess the woman.

SUMMARY:
* All patients fulfilling the selection criteria undergo complete clinical examination and detailed medical history obtained. Each patient had a Case Record Form (CRF) recording participants' name. number, previous deliveries and abortions, age, height, weight, BMI, LMP, past medical and surgical history and contraceptive history.
* All participants will be subjected to transvaginal ultrasound to measure uterine size, endometrial and myometrial thickness, uterine position, cervical length, cervical diameter and for detection of any contraindications for IUD insertion.

Power Doppler Energy (PDE) measurement for subendometrial microvascularization will be done and categorized as women with minor subendometrial vascularization (Classifications I and II) and major subendometrial vascularization (Classifications III, IV and V)

DETAILED DESCRIPTION:
All patients fulfilling the selection criteria undergo complete clinical examination and detailed medical history obtained. Each patient had a Case Record Form (CRF) recording participants' name. number, previous deliveries and abortions, age, height, weight, BMI, LMP, past medical and surgical history and contraceptive history.

- All participants will be subjected to transvaginal ultrasound to measure uterine size, endometrial and myometrial thickness, uterine position, cervical length, cervical diameter and for detection of any contraindications for IUD insertion.

Power Doppler Energy (PDE) measurement for subendometrial microvascularization will be done and categorized as women with minor subendometrial vascularization (Classifications I and II) and major subendometrial vascularization (Classifications III, IV and V)

Only clinicians with proven proficiency in IUD insertion will be allowed to perform insertions.

* Perform a bimanual examination to determine the size, shape, and position of the uterus.
* Insert a warm, moistened speculum.
* Cleanse the cervix with an antiseptic solution.
* Open the sterile insertion instruments without touching the inside of the packet and place within easy reach.
* Remove the tenaculum by its handle and grasp the anterior or posterior lip of the cervix. Close gently to the first notch. Having the woman to cough while the tenaculum is being attached can ease the pinch.
* Apply gentle traction with the tenaculum to straighten the canal.
* Remove the sound by its handle and gently insert it to measure the depth of the uterus. Do not apply great force if there is resistance. Apply further traction to the tenaculum and attempt to re-insert the sound at a different angle. Once the sound is inserted and removed, note the depth of the uterine cavity. The woman can expect to feel cramping as the sound is inserted and withdrawn.
* Open the IUD pack without touching its contents.
* Put on sterile gloves.
* Load the IUD and insert it into the uterine cavity according to the manufacturer instructions. As the IUD is inserted through the cervix into the uterus, the patient may have pain and cramping similar to strong menstrual cramps.
* Gently remove the tenaculum. Tamponade any bleeding from the tenaculum site until it is resolved.
* Trim the strings of the IUD to 3-4 cm in length and note the string length. Avoid cutting the strings too short. If the client or her partner becomes aware of the threads, they may be cut shorter in length at the follow-up visit.
* Remove the speculum and assess the woman.
* Pain score will be assessed using Visual Analogue Scale:

  1. Anticipated pain or current pain before the intervention.
  2. Immediately after speculum insertion.
  3. Immediately after tenaculum placement.
  4. Immediately after uterine sounding.
  5. During or immediately after IUD insertion.
  6. Five minutes after the procedure

     * Follow up at 3 and 6 months to assess women satisfaction with the method, menstrual pattern, symptoms of vaginal/pelvic infection Abdominal pain/tenderness Dyspareunia (woman/partner) Cramping or pregnancy.
     * Vaginal examination to assess any infections or abnormalities and repeat ultrasound examination to assess the position of the IUD

ELIGIBILITY:
Inclusion Criteria:

* Age 20 -41 years
* BMI 18-25 kg/m2
* Women with any parity seeking contraception and choosing IUD as their preferred method after proper and thorough counseling
* Regularly menstruating women (duration of menstruation 3-7 days and length of cycle 22- 35 days).
* Not using any hormonal therapy or anticoagulation

Exclusion Criteria:

* Cervical abnormalities.
* Pregnancy or suspicion of pregnancy
* Congenital or acquired uterine anomalies which distort the uterine cavity (fibroids, endometrial polyps, cervical stenosis, bicornuate uterus, hypoplastic uterus < 6 cm)
* Acute PID or a history of PID within the past 3 months
* Postpartum or post-abortion endometritis within the past 3 months
* Current STI or within the past 3 months (including cervicitis)
* Cervical cancer
* Endometrial cancer
* Malignant gestational trophoblastic disease
* Undiagnosed vaginal bleeding
* Hypersensitivity to any component in the IUD (copper)
* Less than 6 weeks postpartum.
* Neurological or psychological conditions that may affect pain sensation

Ages: 20 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Failed IUD insertion | 9 months
  failure of IUD insertion

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided